CLINICAL TRIAL: NCT03319173
Title: Dietary Ketosis a Metabolic Sister to Calorie Restriction (CR): Fatty Acids Activate AMPK Energy Circuits Modulating Global Methylation Via the SAM/SAH Axis
Brief Title: Dietary Ketosis: Fatty Acids Activate AMPK Energy Circuits Modulating Global Methylation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristlecone Health, Inc. (Industry)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bristlecone-001
Record Dates: First submitted 2017-10-14; First posted 2017-10-24 (Actual); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Mild Cognitive Impairment; Metabolic Syndrome
Keywords: Mild Cognitive Impairment; AMPK activation; DNA global hypo-methylation; Metabolic Syndrome; Ketogenic diet; SAM/SAH Index; S-adenosylmethionine (SAM); S-adenosylhomocysteine (SAH); Region-Specific hyper-methylation; mTOR kinase pathway; AMP/ATP ratio; Low Reduction Potential; High Reduction Potential; Delta G; Exergonic; Endergonic; Epigenetic Histone Modification; Montreal Cognitive Assessment (MoCA); Brief Visual Memory Test-Revised (BVMT-R); Rey Auditory Verbal Learning Task (RAVLT); HOMA-IR
MeSH Terms: conditions — Cognitive Dysfunction; Metabolic Syndrome | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: To assess differences between the control and experimental groups, a mixed model will be fit for each variable separately using both baseline (week 0) and post program (week 12) values for each subject. Models will include week, group, and their interaction as fixed effects, gender as a covariate, and subject as a random effect. To assess significant differences, we will use the difference at week 12 adjusted for the baseline difference, and will report p-values, least squares means, and 95% confidence intervals. Further analysis of treatment effects over time will be examined by comparing the within-group differences over time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Dietary interventions for subjects in the experimental group include clinically regulated meal plans designed to facilitate prolonged benign dietary ketosis (BDK) in order to regulate glucose with restored insulin sensitivity focused at reversing the impaired capacity to switch between fat and carbohydrate oxidation. Subjects will consume 3 meals per day with the following approximate macronutrient breakdown per meal: 65% fat, 25% protein, 10% carbohydrate.
  Both groups will play the Advanced PEAK brain training games on iPhone, iPad or Android devices for 75 minutes per week.
  Interventions: Behavioral: Dietary intervention
- Control group (Active Comparator): Dietary interventions for subjects in the control group include the subjects' current dietary protocol (Standard American Diet-SAD). Subjects will consume 4-6 small meals per day with the following approximate macronutrient breakdown per meal: 50% carbohydrate, 35% protein, 15% fat.
  Both groups will play the Advanced PEAK brain training games on iPhone, iPad or Android devices for 75 minutes per week.
  Interventions: Behavioral: Dietary intervention

INTERVENTIONS:
Behavioral: Dietary intervention — Subjects in the experimental group will receive clinically regulated meal plans designed to facilitate prolonged benign dietary ketosis (BDK) in order to regulate glucose with restored insulin sensitivity focused at reversing the impaired capacity to switch between fat and carbohydrate oxidation.
  Subjects in the control group will follow the their current dietary protocol (Standard American Diet-SAD).

SUMMARY:
The study explores whether selective memory complaints (SMC), mild cognitive impairment (MCI) and the comorbidity of Metabolic Syndrome symptomatic of peripheral and cerebral hypo-metabolism with corresponding epigenetic shifts in global DNA (deoxyribonucleic acid) methylation (away from nutrient availability and toward biosynthesis) are initiated by chronic metabolic inflexibility, over-activation of the mTOR (mammalian target of rapamycin) pathway, and the deregulation of neural oxidative phosphorylation.

DETAILED DESCRIPTION:
Nutritional epigenetics denotes gene-diet interactions and highlights the modulatory role of cellular energy status in aging and age-related diseases like cancer, cardiovascular disease (CVD), diabetes and neurodegeneration. Nutrients are epigenetic modifiers; macro and micronutrients regulate the placement and distribution of DNA histone modifiers distinguishing phenotype from genotype. Cellular energy status (AMP/ATP) modulates the regulatory mechanics of DNA methylation via the SAM (S-adenosylmethionine) methlytransferase and the SAH (S-adenosyl homocysteine) methyltransferase inhibitor index. Whole blood histamine and homocysteine levels provide additional information on the status of methylation. Hyperinsulinemia and cellular insulin resistance dysregulate nutrient sensing pathways; perpetual fed-state signaling exacerbates systemic metabolic inflexibility. Chronic elevations in insulin with long-standing impairments in glucose delivery are associated with profound changes in epigenetic expression consequent of hyper-activation of mTOR and inhibition of AMPK kinase pathways. Dietary ketosis is known to govern adaptive mitonuclear energy availability by increasing cellular reduction potential via >AMP/ATP ratio. AMPK activation adapts rRNA synthesis away from fed-state growth/storage toward energy production/release, common to fasted-states. Research suggests that induced and controlled dietary ketogenesis, a fasting mimetic, transcriptionally modifies gene expression thereby attenuating metabolic diseases.

The study will explore whether early stage memory loss (SMC & MCI) and comorbidity of Metabolic Syndrome are symptomatic of peripheral and cerebral hypo-metabolism resultant of sustained cellular insulin resistance. The investigators will attempt to show that consequent to systemic hyperinsulinemia, mitonuclear crosstalk dysregulates the energy sensing kinases, mTOR/AMPK, thereby modifying the intra/extracellular nutrient signaling pathways. The suppression of AMPK, coupled with chronic fed-state signaling, adapts rRNA synthesis away from nutrient availability toward ATP consuming processes. Increased biosynthesis of proteins, lipids and cholesterol with concurrent inhibition of fat oxidation, energy cofactors (NAD+, SAHH) and programmed apoptosis results in the epigenetic drift of methylation toward global gene activation with region-specific silencing of key regulatory/longevity genes, SIRTs (sirtuins), FOX03 and Nrf2. This global shift in energy is marked by suppression of the SAM/SAH methylation index and correlative jumps in whole blood histamine and/or homocysteine. The study explores whether the aforementioned shift in nutrient sensing pathways modulates metabolic inflexibility via energy shunts toward cytosolic, substrate level phosphorylation via activation of PDK (pyruvate dehydrogenase kinase). An insulin resistant energy surplus (<AMP/ATP) fosters low cellular reduction potential, which triggers mitonuclear crosstalk inhibiting oxidative ATP via PDC (pyruvate dehydrogenase complex), the regulatory gateway between anaerobic glycolysis and oxidative mitochondrial respiration. The study will attempt to show that induced and controlled dietary ketosis initiates the spontaneous/favorable release of energy ( >AMP/ATP), activating the AMPK circuitry thereby inhibiting the synthesis/storage of protein, cholesterol and lipids. Thus, a shift in cellular energy from low reduction potential (ATP/NADH) to high reduction potential (AMP/NAD+) attenuates methylation drift evidenced by marked reductions in biosynthesis: fasting lipid profile (TRI., VLDL, LDL, HDL), LP-IR score (particle concentration/size), HgA1c, fasting insulin, HOMA-IR and epigenetic modification of DNA measured by improved methylation index (>SAM/SAH) with correlating reductions in whole blood histamine and/or homocysteine. The resultant change in cerebral glucose metabolism and correlative improvement in SMC/MCI will be assessed by valid clinical measures of cognition: Montreal Cognitive Assessment (MoCA), Brief Visual Memory Test-Revised (BVMT-R) and Rey Auditory Verbal Learning Task (RAVLT) administered at baseline and weeks 2/4/6/8/10/12.

Research Question: Are selective memory complaints (SMC), mild cognitive impairments (MCI) and comorbid Metabolic Syndrome symptomatic of peripheral/cerebral insulin resistance with a resultant epigenetic drift in methylation away from energy production toward anabolic synthesis/storage, initiated and sustained by metabolic inflexibility, aerobic glycolysis and PDK inhibition of oxidative phosphorylation?

ELIGIBILITY:
Inclusion Criteria:

* Male or Female (age 35-80)
* Previously diagnosed with MetS and/or T2DM as measured by possessing at least two of the following physiological measures: type 2 diabetes, BMI > 30, HgA1c > 5.7%, waist/height ratio > .6, fasting glucose > 125 mg/dL
* Subjective Memory Complaints (SCM) - Subjects score > 3 'yes' answers on the Subjective Memory Complaints Questionnaire
* Previously diagnosed with Mild Cognitive Impairment (MCI)

Exclusion Criteria:

* Previously diagnosed with Alzheimer's disease (AD), dementia or Parkinson's disease

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly J Gibas, Doctorate, Principal Investigator — Bristlecone Health, Inc.
Locations (1):
- Bristlecone Health, Inc., Maple Grove, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Group: Dietary interventions for subjects in the experimental group include clinically regulated meal plans designed to facilitate prolonged benign dietary ketosis (BDK) in order to regulate glucose with restored insulin sensitivity focused at reversing the impaired capacity to switch between fat and carbohydrate oxidation. Subjects will consume 3 meals per day with the following approximate macronutrient breakdown per meal: 65% fat, 25% protein, 10% carbohydrate.
  Both groups will play the Advanced PEAK brain training games on mobile devices for 75 minutes per week.
  Dietary intervention:Subjects in the experimental group will receive clinically regulated meal plans designed to facilitate prolonged benign dietary ketosis (BDK) in order to regulate glucose with restored insulin sensitivity focused at reversing the impaired capacity to switch between fat and carbohydrate oxidation.
  Subjects in the control group will follow the their current dietary protocol (Standard American Diet-SAD).
- Control Group: Dietary interventions for subjects in the control group include the subjects' current dietary protocol (Standard American Diet-SAD). Subjects will consume 4-6 small meals per day with the following approximate macronutrient breakdown per meal: 50% carbohydrate, 35% protein, 15% fat.
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 48 | 50
Completed | 48 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental Group: Dietary interventions for subjects in the experimental group include clinically regulated meal plans designed to facilitate prolonged benign dietary ketosis (BDK) in order to regulate glucose with restored insulin sensitivity focused at reversing the impaired capacity to switch between fat and carbohydrate oxidation. Subjects will consume 3 meals per day with the following approximate macronutrient breakdown per meal: 65% fat, 25% protein, 10% carbohydrate.
  Both groups will play the Advanced PEAK brain training games on iPhone, iPad or Android devices for 75 minutes per week.
  Dietary intervention: Subjects in the experimental group will receive clinically regulated meal plans designed to facilitate prolonged benign dietary ketosis (BDK) in order to regulate glucose with restored insulin sensitivity focused at reversing the impaired capacity to switch between fat and carbohydrate oxidation.
- Control Group: Dietary interventions for subjects in the control group include the subjects' current dietary protocol (Standard American Diet-SAD). Subjects will consume 4-6 small meals per day with the following approximate macronutrient breakdown per meal: 50% carbohydrate, 35% protein, 15% fat.
  Both groups will play the Advanced PEAK brain training games on iPhone, iPad or Android devices for 75 minutes per week.
  Dietary intervention: Subjects in the control group will follow the their current dietary protocol (Standard American Diet-SAD).
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 48 | 50 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 44 | 85
  >=65 years | 7 | 6 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 23 | 25 | 48
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 48 | 50 | 98
MoCA (Montreal Cognitive Assessment) [Least Squares Mean (Inter-Quartile Range); unit: units on a scale] — MoCA score ranges:
  Normal: >= 26; MCI (mild cognitive impairment): 17-25
  units on a scale | 28.38 [27.94 to 28.81] | 20.22 [19.79 to 20.64] | 24.30 [23.50 to 25.1]

OUTCOME MEASURES:

1. Primary Outcome: MoCA (Montreal Cognitive Assessment)
Description: Measures changes in cognitive function over time. Score: 30 points (maximum), 0 points (minimum). Score >25 = normal cognitive function. Score 17-25 = mild cognitive impairment (MCI). Score <17 = increased likelihood of Alzheimer's Disease or dementia.
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Experimental Group; Control Group: MoCA post intervention score
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 48 | 50
score on a scale | 28.38 (0.22) | 20.22 (0.22)
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Other; p < 0.0001, Regression, Linear; Mean Difference (Final Values) = 8.24, 95% CI 2-sided [7.79 to 8.7], Standard Error of Mean 0.23

2. Secondary Outcome: NMR Lipoprofile Particle Size - Small LDL-P
Description: Assessment of changes in Small LDL-P (total small Pattern B)
Time Frame: 12 weeks
Measure: Geometric Least Squares Mean (Standard Error); unit: nmol/L
Groups:
- Experimental Group: Dietary interventions for subjects in the experimental group include clinically regulated meal plans designed to facilitate prolonged benign dietary ketosis (BDK) in order to regulate glucose with restored insulin sensitivity focused at reversing the impaired capacity to switch between fat and carbohydrate oxidation. Subjects will consume 3 meals per day with the following approximate macronutrient breakdown per meal: 65% fat, 25% protein, 10% carbohydrate.
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 48 | 50
nmol/L | 276.24 (29.25) | 588.08 (61.02)
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Other; p < 0.0001, Regression, Linear; Estimate = 0.35, 95% CI 2-sided [0.31 to 0.39], Standard Error of Mean 0.02

3. Secondary Outcome: NMR Lipoprofile Particle Size - LP-IR Score (Lipoprotein Insulin Resistance) Ideal Range: <45
Description: Lipoprotein insulin resistance (LP-IR) is an aggregate score of the 6 lipoprotein parameters range from 0 to 100, with higher scores indicating greater insulin resistance (IR).
Time Frame: 12 weeks
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 48 | 50
score on a scale | 32.13 [28.87 to 35.76] | 50.66 [45.62 to 56.26]
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Other; p < 0.0001, Regression, Linear; Estimate = 0.46, 95% CI 2-sided [0.41 to 0.52], Standard Error of Mean 0.03

4. Secondary Outcome: Fasting Triglycerides
Description: Assessment of changes in fasting triglycerides over time. Ranges: < 150 mg/dL
Time Frame: 12 weeks
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 48 | 50
mg/dL | 87.23 [76.58 to 99.35] | 131.73 [115.96 to 149.64]
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Other; p < 0.0001, Regression, Linear; Estimate = 0.514, 95% CI 2-sided [0.47 to 0.56], Standard Error of Mean 0.02

5. Secondary Outcome: Triglyceride/HDL Ratio
Description: Assessment of changes in Triglyceride/HDL ratio over time.
Time Frame: 12 weeks
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 48 | 50
ratio | 1.67 [1.41 to 1.99] | 2.69 [2.28 to 3.19]
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Other; p < 0.0001, Regression, Linear; Estimate = 0.44, 95% CI 2-sided [0.40 to 0.49], Standard Error of Mean 0.02

6. Secondary Outcome: Fasting Insulin
Description: Assessment of changes in fasting insulin over time. Ranges: < 2.6-11.1 mU/L
Time Frame: 12-weeks
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mU/L
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 48 | 50
mU/L | 7.32 [6.37 to 8.42] | 11.25 [9.81 to 12.91]
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Other; p < 0.0001, Estimate; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [0.40 to 0.49], Standard Error of Mean 0.02

7. Secondary Outcome: Fasting Glucose
Description: Assessment of changes in fasting glucose over time. Ranges: < 74-100 mg/dL
Time Frame: 12-weeks
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 48 | 50
mg/dL | 85.9 [82.64 to 89.30] | 109.61 [105.52 to 113.85]
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Other; p < 0.0001, Regression, Linear; Estimate = 0.75, 95% CI 2-sided [0.72 to 0.78], Standard Error of Mean 0.01

8. Secondary Outcome: HOMA-IR
Description: Assessment of changes in HOMA-IR (Homeostatic Model Assessment of Insulin Resistance) over time. Ranges: < 1.0
Time Frame: 12-weeks
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 48 | 50
units on a scale | 1.55 [1.32 to 1.83] | 3.05 [2.60 to 3.57]
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Other; p < 0.0001, Estimate; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [0.30 to 0.37], Standard Error of Mean 0.02

9. Secondary Outcome: HgA1c
Description: Assessment of changes in HgA1c (Hemoglobin A1c) over time.
Time Frame: 12-weeks
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: percentage of glycated hemoglobin
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 48 | 50
percentage of glycated hemoglobin | 5.19 [5.11 to 5.28] | 5.82 [5.73 to 5.91]
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Other; p < 0.0001, Regression, Linear; Estimate = 0.87, 95% CI 2-sided [0.85 to 0.88], Standard Error of Mean 0.01

10. Secondary Outcome: Weight
Description: Assessment of changes in weight over time as measured in pounds.
Time Frame: 12-weeks
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: pounds
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 48 | 50
pounds | 200.23 [189.46 to 211.62] | 210.60 [199.49 to 222.32]
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Other; p < 0.0001, Regression, Linear; Estimate = 0.87, 95% CI 2-sided [0.85 to 0.88], Standard Error of Mean 0.01

11. Secondary Outcome: Body Fat Mass (BFM)
Description: Assessment of changes in body fat mass over time as measured in pounds.
Time Frame: 12-weeks
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: pounds
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 48 | 50
pounds | 67.95 [62.21 to 74.21] | 79.35 [72.78 to 86.52]
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Other; p < 0.0001, Regression, Linear; Estimate = 0.75, 95% CI 2-sided [0.71 to 0.80], Standard Error of Mean 0.02

12. Secondary Outcome: VLDL
Description: Assessment of changes in VLDL (very low density lipoprotein carrier) over time. Ranges: < 5-40 mg/dL
Time Frame: 12-weeks
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 48 | 50
mg/dL | 17.45 [15.32 to 19.87] | 26.35 [23.19 to 29.93]
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Other; p < 0.0001, Regression, Linear; Estimate = 0.51, 95% CI 2-sided [0.47 to 0.56], Standard Error of Mean 0.02

13. Secondary Outcome: SAM/SAH Ratio (S-adenosylmethionine/S-adenosylhomocysteine)
Description: Assessment of changes in SAM/SAH (S-adenosylmethionine/S-adenosylhomocysteine) ratio Range: >4.0
Time Frame: 12-weeks
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 48 | 50
ratio | 4.938 [4.538 to 5.372] | 4.491 [4.119 to 4.896]
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Other; p < 0.0001, Regression, Linear; Estimate = 1.130, 95% CI 2-sided [1.104 to 1.156], Standard Error of Mean 0.013

14. Secondary Outcome: SAM (S-adenosylmethionine)
Description: Assessment of changes in SAM (S-adenosylmethionine)
Time Frame: 12-weeks
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 48 | 50
nmol/L | 89.784 [84.767 to 95.099] | 88.177 [83.131 to 93.529]
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Other; p < 0.0001, Regression, Linear; Estimate = 1.037, 95% CI 2-sided [1.025 to 1.049]

15. Secondary Outcome: SAH (S-adenosylhomocysteine)
Description: Assessment of changes in SAH (S-adenosylhomocysteine) Range: 10-22 nmol/L
Time Frame: 12-weeks
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 48 | 50
nmol/L | 18.257 [17.685 to 18.847] | 19.566 [18.938 to 20.214]
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Other; p < 0.0001, Regression, Linear; Estimate = 0.93, 95% CI 2-sided [0.91 to 0.94], Standard Error of Mean 0.008

16. Secondary Outcome: Adenosine
Description: Assessment of changes in Adenosine Range: 20-80 nmol/L
Time Frame: 12-weeks
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 48 | 50
nmol/L | 23.363 [22.413 to 24.352] | 21.475 [20.581 to 22.407]
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Other; p < 0.0001, Regression, Linear; Estimate = 1.122, 95% CI 2-sided [1.096 to 1.149], Standard Error of Mean 0.014

ADVERSE EVENTS:
Time Frame: 12-weeks
Description: Study protocol/procedures non-invasive
Groups:
- Control Group: Dietary interventions for subjects in the control group include the subjects' current dietary protocol (Standard American Diet-SAD). Subjects will consume 4-6 small meals per day with the following approximate macronutrient breakdown per meal: 50% carbohydrate, 35% protein, 15% fat.
  Both groups will play the Advanced PEAK brain training games on iPhone, iPad or Android devices for 75 minutes per week.
  Subjects in the control group will follow the their current dietary protocol (Standard American Diet-SAD).
Arm/Group | Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/50
Other Adverse Events (participants affected / at risk) | 0/48 | 0/50

LIMITATIONS AND CAVEATS:
No limitations or caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT03319173/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT03319173/SAP_001.pdf